CLINICAL TRIAL: NCT00582374
Title: Periodontal Disease, Inflammatory Markers, and Preterm Birth
Brief Title: Periodontal Disease and Preterm Birth
Status: Withdrawn | Type: Observational
Why Stopped: PI passed away unexpectedly
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: PeriodontalPreTermBirth
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Periodontal Disease; Preterm Birth; Low Birth Weight
Keywords: Periodontal Disease; Preterm Birth; Low Birth Weight; Pregnancy
MeSH Terms: conditions — Periodontal Diseases; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Gingival crevicular fluid (GCF) and Vaginal Fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Pregnant Women

SUMMARY:
To determine the relationship between periodontal disease and upper genital tract inflammation in pregnancy. To determine whether certain fluid levels in the oral cavity and the vagina are associated with preterm birth or low-birth weight.

DETAILED DESCRIPTION:
Patients will be enrolled in the study at their first prenatal visit after the details of the study have been discussed. Potential subjects will be presented with a questionnaire to determine eligibility for the study. The patient will be scheduled for an exam between 18-24 weeks at which time they will undergo a periodontal assessment, to determine the presence or absence of periodontal disease, a sampling of gingival crevicular fluid (GCF) and a vaginal swab collection. Periodontal disease will be determined by measuring the depth of gingival sulci, amount of periodontal attachment loss, and prevalence of gingival bleeding at six sites for each tooth present.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 15-35
* Singleton gestation

Exclusion Criteria:

* Diabetes prior to pregnancy
* Require antibiotic prophylaxis prior to dental treatment
* Require steroids during pregnancy

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant women from the OU Medical Center Women's Clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-03; Primary Completion 2009-03 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
To determine the relationship between periodontal disease and upper genital tract inflammation as measured by cytokine levels IL-6, IL-1, and TNF-α and MMP levels from the posterior fornix of the vagina. | 4 years

SECONDARY OUTCOMES:
To determine whether IL-1β levels in the oral cavity and the vagina are associated with preterm birth or low-birth weight. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric Knudtson, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States